CLINICAL TRIAL: NCT04221828
Title: Phase 2 Trial of NanoPac Focal Therapy for Prostate Cancer in Subjects Undergoing Radical Prostatectomy
Brief Title: Trial of NanoPac Focal Therapy for Prostate Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of enrollment
Sponsor: NanOlogy, LLC (Industry)
Collaborators: US Biotest, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NANOPAC-2019-01
Expanded Access: NCT03756311 (No longer available)
Record Dates: First submitted 2020-01-07; First posted 2020-01-09 (Actual); Results first posted 2022-03-29 (Actual); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Prostate Cancer; Prostate Adenocarcinoma; Prostate Cancer Adenocarcinoma; Prostatic Neoplasm; Urogenital Neoplasms; Genital Neoplasms, Male; Localized Cancer
Keywords: paclitaxel
MeSH Terms: conditions — Prostatic Neoplasms; Urogenital Neoplasms; Genital Neoplasms, Male | interventions — Powders; Suspensions; Paclitaxel

STUDY DESIGN:
Intervention Model Description: Open-label, single group, safety, efficacy, and pharmacokinetic study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- NanoPac (Experimental): Direct injection of NanoPac at 15 mg/mL at a volume not to exceed the volume of the prostate cancer lesion (no more than 10% of total prostate volume). NanoPac will be administered on up to three occasions, with at least 28 days between each dose.
  Interventions: Drug: NanoPac (sterile nanoparticulate paclitaxel) Powder for Suspension

INTERVENTIONS:
Drug: NanoPac (sterile nanoparticulate paclitaxel) Powder for Suspension — NanoPac is manufactured using a Precipitation with Compressed Antisolvent (PCA) technique that employs supercritical carbon dioxide and acetone to generate paclitaxel nanoparticles. For clinical administration, the NanoPac powder in vial is suspended with Sterile Reconstitution Solution (1% Polysorbate 80, NF in 0.9% Sodium Chloride for Injection, USP) and then further diluted with 0.9% Sodium Chloride for Injection, USP, to achieve the final clinical formulation.
  Other Names: paclitaxel

SUMMARY:
This study evaluates the use of NanoPac injected directly into the prostate lesion in men with prostate cancer.

DETAILED DESCRIPTION:
NanoPac is very small (submicron) particles of the chemotherapy drug, paclitaxel, which is administered intravenously in a number of types of cancer. These submicron particles are injected directly into solid tumors to target cancer at the site of disease with less systemic exposure than intravenously administered chemotherapy. In this study, this submicron particle paclitaxel will be injected directly into the prostate lesion in men with prostate cancer scheduled for prostatectomy on up to three different occasions. All subjects in the study will receive NanoPac and will be evaluated to see if NanoPac is safe, well-tolerated, and has an impact on prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age;
* Histopathologically proven adenocarcinoma of the prostate:

  * Localized cancer;
  * Subjects with tumors classified as <T3 per TNM classification, Gleason score≥ 6;
* Prostate tumor must be able to be visualized on mpMRI;
* Already considered to be candidate for radical prostatectomy;
* Considered appropriate for treatment with paclitaxel therapy;
* Laboratory requirements:

  * WBC >2500/mm3
  * Neutrophil >1500/mm3
  * Hemoglobin >10 mg/dL
  * Platelet >100,000/ mm3
  * AST and ALT <2.5 x ULN
  * Total bilirubin <1.5 x ULN
  * Calculated creatinine clearance ≥ 30 ml/min
  * Normal PT/INR and PTT;
* ECOG of 0 or 1;
* International Prostate Symptom Score (I-PSS) less than or equal to 20;
* If sexually active, willing to use double condoms from time of NanoPac injection until prostatectomy;
* Agree to all study procedures and provide signed informed consent;

Exclusion Criteria:

* Evidence of locally advanced or metastatic disease;
* Prostate size ≥ 50 cc;
* Prior prostatectomy, including surgery for any benign condition (such as TURP);
* Anticipated use of concomitant chemotherapy (other than the protocol specified agents), immunotherapy, or systemic use of hormonal therapy (such as GnRH analogs, antiandrogens, androgen receptor inhibitors, and 5-α reductase inhibitors) while on study prior to surgery;
* Treatment with a prior investigational medication within 30 days of first dose of study agent;
* Any previous local treatment of the prostate (e.g. radiation, HIFU, cryotherapy, Focal Irreversible Electroporation, Photodynamic Therapy, Laser Induced Thermometry);
* Any other condition (e.g., psychiatric disorder) that, in the opinion of the Investigator, may interfere with the subject's ability to comply with the study requirements or visit schedule;
* Known sensitivity to any of the study agent components;
* History of prior malignancy that has not been in remission for >5 years, with the exception of basal cell or squamous cell carcinoma.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2020-10-20 (Actual); Primary Completion 2021-01-27 (Actual); Study Completion 2021-02-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shelagh Verco, PhD, Study Director — US Biotest, Inc.
Locations (4):
- United States (4):
  - Moffitt Cancer Center, Tampa, Florida
  - University of Kansas Medical Center, Kansas City, Kansas
  - Henry Ford Health System, Detroit, Michigan
  - University of Missouri, Columbia, Missouri

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | NanoPac
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | NanoPac
Number analyzed (Participants) | 1
Age, Continuous [Mean (Full Range); unit: years] | 56 [56 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 1
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
PSA [Number; unit: ng/mL] | 5.4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment Emergent Adverse Events
Description: Treatment emergent adverse events (including changes in laboratory assessments, physical examination findings, and vital signs)
Time Frame: Day 1 to Day 85
Measure: Count of Participants; unit: Participants
Arm/Group | NanoPac
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Tumor Response Based on Histologic Evaluation of Biopsied Prostate Samples (Gleason Score)
Description: Prostate tissue samples obtained from a biopsy performed prior to baseline and prostatectomy. Histologic evaluation of these samples will be used to determine the Gleason score, and the results at baseline and Day 92 will be used to evaluate the tumor response to NanoPac. The Gleason score is calculated by adding together the two grades of cancer cells that make up the largest areas of the biopsied tissue sample. The Gleason score usually ranges from 6 to 10. The lower the Gleason score, the more the cancer cells look like normal cells and are likely to grow and spread slowly; a higher Gleason score is likely to indicate a worse outcome. The Gleason score is used to help plan treatment and determine prognosis.
Time Frame: Up to 2 weeks prior to Day 1 and Day 92
Population: Data not collected
Arm/Group | NanoPac
Number analyzed (Participants) | 0

3. Secondary Outcome: Tumor Response Based on Change in Percentage of Sample Considered Adenocarcinoma
Description: Tissues excised from the dominant lesion during prostatectomy (Day 92) will be evaluated for the percentage considered adenocarcinoma and compared to biopsy sample obtained at baseline.
Time Frame: Up to 2 weeks prior to Day 1 and Day 92
Population: Data not collected
Arm/Group | NanoPac
Number analyzed (Participants) | 0

4. Secondary Outcome: Tumor Invasion Into Surrounding Tissues
Description: The proportion of subjects with local invasion as measured by mpMRI at the final study visit will be compared to screening (baseline)
Time Frame: Up to 1 month prior to Consent and Day 85
Population: Data not collected
Arm/Group | NanoPac
Number analyzed (Participants) | 0

5. Secondary Outcome: Tumor Response Based on Change in Image Volume on mpMRI
Description: Tumor response to treatment with NanoPac will be determined by evaluating the change in image volume with multiparametric MRI (mpMRI) obtained prior to consent and again at the final study visit.
Time Frame: Up to 1 month prior to Consent and Day 85
Population: Data not collected
Arm/Group | NanoPac
Number analyzed (Participants) | 0

6. Secondary Outcome: Change in PSA Density
Description: PSA density (PSAD), is a calculation of the serum PSA level divided by the volume of the prostate gland. PSA density has been used as a prognostication tool in helping decide treatment approach. PSA density measured at the final study visit will be compared to screening (baseline)
Time Frame: Up to 2 weeks prior to Day 1 and Day 85
Measure: Number; unit: percent change in PSAD
Arm/Group | NanoPac
Number analyzed (Participants) | 1
percent change in PSAD | 0

7. Secondary Outcome: Change in PI-RADS Score
Description: The Prostate Imaging Reporting and Data System (PI-RADS) assessment uses a five-point scale based on the probability that a combination of mpMRI findings on T2 weighting (T2W), Diffusion Weighted Imaging (DWI), and Dynamic Contrast Enhancement (DCE) correlates with the presence of a clinically significant cancer in the prostate gland. A PI-RADS score of 1 is considered to be most probably benign and a score of 5 is considered to be highly suspicious of prostate malignancy. PI-RADS score will be measured at screening (baseline) and at the final study visit.
Time Frame: Up to 2 weeks prior to Day 1 and Day 85
Population: Data not collected
Arm/Group | NanoPac
Number analyzed (Participants) | 0

8. Secondary Outcome: Effect on Tumor Presence in Lymph Nodes
Description: Optional PSMA PET scan performed prior to first NanoPac injection and prior to prostatectomy
Time Frame: Up to 2 weeks prior to Day 1 and Day 92
Population: Data not collected
Arm/Group | NanoPac
Number analyzed (Participants) | 0

9. Secondary Outcome: Concentration of Paclitaxel in the Systemic Circulation Post-injection
Description: Pharmacokinetic samples will be obtained on days of NanoPac injection and other clinic visits.
Time Frame: Days 1, 8, 15, 29, 36, 43, 50, 57, 64, 71, and 85
Population: Data not collected
Arm/Group | NanoPac
Number analyzed (Participants) | 0

10. Secondary Outcome: Presence or Absence of Paclitaxel in Ejaculate
Description: Ejaculate samples will be collected for analysis of the presence or absence of paclitaxel.
Time Frame: Days 15, 43, 57, and 85
Population: Data not collected
Arm/Group | NanoPac
Number analyzed (Participants) | 0

11. Secondary Outcome: Presence or Absence of Paclitaxel in Tissues Obtained at Prostatectomy
Description: At the time of prostatectomy, available tissues including the tumor, the ipsilateral lobe of the prostate, the contralateral lobe of the prostate, and pelvic lymph nodes, will be evaluated for the presence or absence of paclitaxel
Time Frame: Day 92
Population: Data not collected
Arm/Group | NanoPac
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Day 1 to Day 85
Arm/Group | NanoPac
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

LIMITATIONS AND CAVEATS:
Study was terminated early due to lack of enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-09-08): https://cdn.clinicaltrials.gov/large-docs/28/NCT04221828/Prot_SAP_001.pdf